CLINICAL TRIAL: NCT00145587
Title: Allogeneic Hematopoietic Stem Cell Transplantation for Children Affected With Malignant Osteopetrosis: A Pilot Study
Brief Title: Stem Cell Transplantation for Children Affected With Osteopetrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the principal investigator having left the institution.
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPBMT2
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Results first posted 2011-08-22 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2011-01

CONDITIONS: Osteopetrosis
Keywords: Osteopetrosis; Autosomal recessive bone disease; Haploidentical stem cell transplantation; Allogeneic stem cell transplantation; T-cell depletion methodology; Miltenyi Biotec CliniMACS stem cell selection device
MeSH Terms: conditions — Osteopetrosis | interventions — Stem Cell Transplantation; Antibodies; Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Stem Cell Transplantation; Device: Miltenyi Biotec CliniMACS; Drug: Systemic chemotherapy and antibodies

INTERVENTIONS:
Procedure: Stem Cell Transplantation — An infusion of HLA partially matched family member donor stem cells processed through the use of the investigational Miltenyi Biotec CliniMACS device.
  Other Names: Haploidentical stem cell transplant; Allogeneic stem cell transplant
Device: Miltenyi Biotec CliniMACS — Stem cell selection device
  Other Names: T-cell depletion
Drug: Systemic chemotherapy and antibodies — Haploidentical stem cell transplant recipients will receive a reduced intensity conditioning regimen consisting of OKT-3, Fludarabine, Thiotepa , and Melphalan followed by an infusion of a T-cell depleted donor stem cell product. Rituximab will be administered within 24 hours of the infusion in an effort to prevent post transplantation lymphoproliferative disorders (PTLPD). In addition to T-cell depletion of the donor product, cyclosporine will be provided as prophylaxis for (GVHD)Graft versus Host Disease
  Recipients of a matched sibling donor product will receive a myeloablative conditioning regimen consisting of busulfan and cyclophosphamide. Cyclosporine will be administered for GVHD prophylaxis.
  Other Names: Transplantation for Osteopetrosis

SUMMARY:
Malignant infantile osteopetrosis (MIOP) is a rare fatal genetic disorder that is characterized by the bone's inability to regulate remodeling. The only curative therapy is hematopoietic stem cell transplantation. Stem cells provided from an HLA identical matched sibling donor is the standard of care, but not feasible for the majority of patients. In addition, due to the potentially rapid progression of this disease, the time to identify a suitable HLA matched unrelated donor is not optimal. Therefore this study is designed to test the hypothesis that children with osteopetrosis can properly engraft hematopoietic stem cells that are donated from a partially matched parental donor, or "haploidentical" stem cell donor that are processed on the investigational device, CliniMACS selection system.

DETAILED DESCRIPTION:
The primary objective of this trial will be answered strictly by those patients enrolled who receive a haploidentical stem cell donor graft.

Patients with a matched sibling donor will be offered participation in this clinical trial and will receive a standard myeloablative conditioning regimen followed by the infusion of an unmanipulated bone marrow graft. However, data from these transplant recipients will be reported in a descriptive manner only.

Secondary Objectives in this trial include the following:

* To describe the outcome of children with MIOP who receive hematopoietic stem cells from a matched sibling donor or a haploidentical donor utilizing a uniform approach one year from transplant
* To estimate the fraction of children with MIOP who have a genetic defect correlating to the osteopetrosis phenotype
* To assess carrier-state of the genetic mutation in parents with an affected child
* To assess carrier-state of the genetic mutation in siblings of affected children
* To estimate the effect of age at the time of hematopoietic stem cell transplantation on the overall outcome of children with MIOP
* To describe the kinetics of select cytokine expression before and after transplantation

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignant osteopetrosis as documented by bone marrow biopsy and radiographic imaging
* A suitable hematopoietic stem cell donor is available

Exclusion Criteria:

* Participant has the Carbonic Anhydrase II (CAII) deficiency osteopetrosis variant
* Symptomatic cardiac disease or evidence of significant cardiac dysfunction by ECHO (shortening fraction <30%)
* Creatinine clearance ≤ 40ml/min/1.73m^2
* Bilirubin ≥ 3mg/dL
* SGPT ≥ 500 U/L
* Evidence of current severe infection which would preclude ablative chemotherapy or a successful transplantation
* Karnofsky or Lansky score < 70 noting expected abnormalities

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-07; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Kasow, DO, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: OPBMT2 was activated, July 2004. From September, 2004 through February, 2008, six transplant participants, five donors, and four genetic testing participants were recruited and enrolled on the study.
Pre-assignment Details: Of the fifteen enrollments, the donors and genetic-testing participants did not receive transplants. Of the six transplant participants, five where eligible for and received a haploidentical hematopoietic stem cell transplant (HSCT) and one received a sibling donor HSCT.
Groups:
- Haplo: Patients to receive a haploidentical hematopoietic stem cell transplantation (HSCT).
- Sibling: Genetic testing
Period: Overall Study
Arm/Group | Haplo | Sibling
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haplo | Sibling | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 1 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Engraftment
Description: To determine the need for blood or platelet transfusions and the presence of donor cells being present in the transplant recipient's bone marrow or peripheral blood by 100 day after transplantation for children with malignant infantile osteopetrosis who have received a haploidentical stem cell graft.
Time Frame: 100 days post-transplant
Population: From September 2004 to March 2009, 5 consecutive MIOP patients were treated using mismatched family member donors. Favorable engraftment refers to the transplant patient not requiring blood or platelet transfusions and the presence of donor cells being present in the transplant recipient's bone marrow or peripheral blood.
Measure: Number; unit: Participants
Arm/Group | Haplo | Sibling
Number analyzed (Participants) | 5 | 1
Participants
  Favorable engraftment | 5 | 1
  Un-favorable engraftment | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from September, 2004 through February, 2008.
Arm/Group | Haplo | Sibling
Serious Adverse Events (participants affected / at risk) | 5/5 | 1/1
Other Adverse Events (participants affected / at risk) | 5/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haplo (N=5) | Sibling (N=1)
Fever without Neutropenia (General disorders) | 2 (4) | 0 (0)
Delayed gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, Diffuse Alveolar (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infection, CMV Pneumonitis (Infections and infestations) | 1 (1) | 0 (0)
Infection, Moraxella Catarrhalis, Upper Respiratory (Infections and infestations) | 1 (1) | 0 (0)
Infection, Respiratory Syncytial Virus (Infections and infestations) | 1 (1) | 0 (0)
Infection, Rotavirus, Stool (Infections and infestations) | 1 (1) | 0 (0)
Infection, Staph Aureus, Tracheostomy Site (Infections and infestations) | 1 (1) | 0 (0)
Adult Respiratory Distress Syndrome Related To Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration Pneumonia Related to Tracheal Bleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Infection, Methicillin Resistant Staphylococcus Aureus Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haplo (N=5) | Sibling (N=1)
Allergic Drug Reaction, OKT3 (Immune system disorders) | 3 (3) | 0 (0)
Allergic Drug Reaction, Vancomycin (Immune system disorders) | 1 (1) | 0 (0)
Allergic Reaction, Platelet Transfusion (Immune system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Secondary Graft Failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia, Asymptomatic (Cardiac disorders) | 1 (1) | 0 (0)
Prolonged QT interval (Cardiac disorders) | 0 (0) | 1 (1)
Edema, Lower Extremity (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 4 (5) | 1 (1)
Hypotension (Cardiac disorders) | 2 (3) | 1 (1)
Pulmonary Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Fever without Neutropenia (General disorders) | 3 (6) | 1 (2)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Graft Versus Host Disease (GVHD), Chronic, Skin; Limited/ (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash, Generalized (Skin and subcutaneous tissue disorders) | 4 (7) | 0 (0)
Transient Erythematous Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
GI Reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1)
Bilateral Subdural Hematomas (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding from ear (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Bleeding, Multisite: Oral, Nasal, Hickman Line Site (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bleeding, Tracheal Granuloma (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hematemesis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Petechiae (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Elevated GGT (Hepatobiliary disorders) | 1 (1) | 1 (2)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Hepatobiliary disorders) | 1 (1) | 1 (2)
SGOT Measurement, Abnormal Level (Hepatobiliary disorders) | 2 (3) | 1 (1)
SGPT Measurement, Abnormal Level (Hepatobiliary disorders) | 2 (3) | 1 (1)
Veno-occlusive disease of the liver (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infection, Adenovirus, Stool (Infections and infestations) | 0 (0) | 1 (1)
Infection, Adenovirus, Tracheal Aspirate (Infections and infestations) | 0 (0) | 1 (1)
Infection, Aspergillus, Endotracheal Tube (Infections and infestations) | 0 (0) | 1 (1)
Febrile Neutropenia (Infections and infestations) | 3 (4) | 0 (0)
Infection, Bacillus, Hickman Line (Infections and infestations) | 1 (1) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 2 (2) | 0 (0)
Infection, Coagulase Negative Staphylococcus, Hickman Line Site (Infections and infestations) | 1 (2) | 0 (0)
Infection, Coagulase Negative Staphylococcus, Tracheostomy (Infections and infestations) | 0 (0) | 1 (1)
Infection, Cytomegalovirus, Tracheal Aspirate (Infections and infestations) | 1 (1) | 1 (1)
Infection, Enterococcus Faecalis, Urinary Tract (Infections and infestations) | 1 (1) | 0 (0)
Infection, Haemophilus Influenzae, Tracheal Aspirate (Infections and infestations) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (4) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Twitching/Staring Episode (Nervous system disorders) | 1 (1) | 0 (0)
Otalgia (General disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Infiltrates, Pulmonary (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nephromegaly (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Insufficiency (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Graft Versus Host Disease (GVHD), Acute, Skin; Maximum Stage 3, Overall Grade 2 (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hematuria (Blood and lymphatic system disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
This study closed prior to completion of enrollment due to the principal investigator having left the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes